CLINICAL TRIAL: NCT05283577
Title: Electroacupuncture for the Management of Symptom Clusters in Cancer Patients and Survivors (EAST): A Feasibility Study
Brief Title: Electroacupuncture for the Management of Symptom Clusters in Cancer Patients and Survivors
Acronym: EAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Founding Chair and Professor of Clinical Pharmacy, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20216732
Record Dates: First submitted 2022-02-03; First posted 2022-03-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: This is a randomized sham-controlled, patient and assessor-blinded pilot trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Each participant will attend a total of 10 treatment visits (one visit per week), over the course of 10 weeks. Each EA session will be approximately 1 hour. Participants in the treatment arm will receive EA at 13 standardized acu-points that were chosen for their therapeutic effects.
  Interventions: Other: Electroacupuncture
- Control Arm (Sham Comparator): Each participant in the control arm will attend a total of 10 treatment visits (one visit per week), over the course of 10 weeks. Participants in the control arm will receive electrical stimulation at non-disease related acu-points for approximately 1 hour per session.
  Interventions: Other: Sham-Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — EA at 13 standardized acu-points that were chosen for their therapeutic effects: Shenting (GV24), Baihui (DU20), Sinshencong (EX-HN1), Zhongwan (CV12), Guanyuan (CV4), Neiguan (PC6) bilateral, Shenmen (HT7) bilateral, Zusanli (ST36) bilateral, Sanyinjiao (SP6) bilateral, Taixi (KI3) bilateral, Zhaohai (KI6) bilateral, Hegu (LI4) bilateral, Taichong (LIV3) bilateral
  Arms: Treatment Arm
Other: Sham-Electroacupuncture — Non-disease related points with electrical stimulation: Pianli (LI6) bilateral, Wenliu (LI7) bilateral, Fuyang (BL59) bilateral, Kunlun (BL60) bilateral, Sanyangluo (TE8), Sidu (TE9) bilateral, Daheng (SP15) bilateral
  Arms: Control Arm

SUMMARY:
This is a sham-controlled, patient and assessor-blinded pilot trial to evaluate the feasibility of administering EA as an intervention for symptom clusters in cancer patients and survivors, and to evaluate the degree that EA could reduce symptom clusters and the possible underlying mechanisms through examining its influence on biomarkers that are linked with the symptoms.

Participants will be randomized to either the treatment arm (those who will receive EA) or the control arm (those who will receive sham-EA). The treatment period for both groups will be 10 weeks. There will be one study visit a week over the course of the 10-week treatment period, for a total of 10 study treatment visits. Participants in the treatment arm will receive EA at 13 standardized acu-points that have been chosen for their therapeutic effects. Participants in the control arm will receive electrical stimulation at non-disease acu-points. There will be four data collection time points for each participant: (1) baseline, (2) mid-treatment (5 weeks from baseline), (3) end of treatment (10 weeks from baseline), and (4) 4 weeks after end of treatment (14 weeks from baseline). At each of these timepoints, 10mL of peripheral blood will be collected for a biomarker analysis and participants will be asked to complete 4 questionnaires and a computerized cognitive test to evaluate their cognitive function, fatigue level, insomnia, psychological distress, and quality of life. An optional neuroimaging procedure will be available to all eligible participants. In total, study participation will last for 14 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy, safety, and feasibility of offering electroacupuncture as an intervention to improve cancer-related symptoms (cognitive impairment, fatigue, psychological distress and insomnia) and quality of life among cancer patients and survivors receiving care at UCI Health. In addition, changes in biomarkers (plasma BDNF, pro-inflammatory cytokines and mitochondrial DNA) known to be associated with cancer-related symptoms. We hypothesize that EA is an effective, safe, and feasible intervention for cancer patients and survivors.

Our specific aims are as follows:

* To compare the efficacy of EA versus sham-EA control in reducing cognitive toxicity, fatigue, psychological distress, insomnia, and to improve quality of life.
* To evaluate the impact of EA versus sham-EA control on biomarkers, including circulating BDNF, pro-inflammatory cytokines (IL-1β, IL-4, IL-6, IL-8, IL-10, TNF-alpha), mitochondrial DNA (oxidative stress indicator).
* To compare the reduction of structural (brain gray matter) and functional connectivity at the prefrontal, medial temporal, and parietal brain regions pre- and post-EA treatment.
* To assess the safety and feasibility of administering EA to manage symptom clusters in cancer patients and survivors.
* As the UCI MINDS C2C registry (UCI IRB Approval #: HS# 2015-2494) will be leveraged to recruit some patients, we will quantify the characteristics associated with non-response to our study advertisement among C2C registrants using C2C-collected data.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer that have received anti-cancer treatment
* 16 years of age or older
* Life expectancy ≥ 6 months
* Complaints of one or more of the following symptoms: memory impairment/attention deficit, fatigue, insomnia, depression, or anxiety over the past 7 days

Exclusion Criteria:

* Presence of metastasis
* Severe needle phobia
* Severe psychiatric or medical disorders which would affect cognitive assessments
* Known bleeding disorder (e.g. hemophilia, Von Willebrand's disease, thrombocytopenia)
* Has pacemaker or other electronic metal implants
* Epilepsy
* Already receiving acupuncture therapy or received acupuncture treatment in the past 3 months.
* Breastfeeding, pregnant or are planning get pregnant during the study period

Additional exclusion criteria for optional neuroimaging procedure:

- Has any contraindications to fMRI including metal fragments/implants in the body, sever claustrophobia, and non-removable metal orthodontic braces, metallic retainers and oral wires.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Cognitive Function (FACT-Cog version 3) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  All subjects will complete the FACT-Cog version 3 questionnaire to assess self-perceived subjective cognitive function. FACT-Cog is a validated questionnaire containing 33 items in the domains of concentration, functional interference, mental acuity, memory, multitasking and verbal fluency. Total score is calculated by summing scores from all the items and ranges from 0-148, and higher scores represent better subjective cognitive functioning.

SECONDARY OUTCOMES:
Objective Cognitive Function (CANTAB®,) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  All subjects will complete Cambridge Neuropsychological Test Automated Battery (CANTAB®), to assess objective cognitive functions. CANTAB® is a computerized cognitive testing software to assess various cognitive domains. Both subjective and objective assessments are recommended by the International Cognition and Cancer Task Force (ICCTF).
Fatigue (MFSI-SF) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  Multidimensional Fatigue Symptom Inventory- Short Form (MFSI-SF) is a validated questionnaire that comprises of 30 items and contains 5 subscales, each with 6 items: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor. The total score is obtained by subtracting the vigour subscale from the sum of all the dimensions (total score range from 24 to 96), with a higher score indicating higher fatigue level.
Psychological Distress and Insomnia (RSCL) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  The Rotterdam Symptom Checklist (RSCL) will be used to measure the psychological symptoms (anxiety and depression) and insomnia. Psychological distress is indicated by a score of >16 in the psychological domain (range 7 to 28). Insomnia is measured by a single item in the checklist (not at all, a little, quite a bit, very much).
Quality of Life (EORTC QLQ-30) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-30) is a validated questionnaire developed to assess cancer patients' health-related quality of life. It incorporates 5 functional scales (cognitive, emotional, physical, role, and social), symptom scales (e.g. pain, fatigue, insomnia), and a global health scale. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale. Higher scores represent a better global health status and better degree of functioning while lower symptom scores indicate less severe symptoms.
Quality of Life (EQ-5D-5L) | All the mean scores will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The mean score changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  EQ-5D comprises a visual analog scale of general health status ranging from 0 (worst imaginable) to 100 (best imaginable) and a descriptive system based on five dimensions of health status: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D descriptive index responses were mapped into a single dimension health utility index (UI) ranging from death (0) to full health (1), with health states worse than death being possible (<0), by using utility weights for the US population.
Safety Monitoring | Through study completion, an average of 14 weeks per participant.
  Participants will be monitored for adverse events such as bruising, pain or discomfort, bleeding and possible infections. Severity are graded according to the Common Terminology Criteria for Adverse Events V5.
Biomarkers - Plasma BDNF (pg/ml) | BDNF levels will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  Plasma brain-derived neurotropic factor (BDNF) levels at each time point, and changes from baseline
Biomarkers - Plasma cytokines (IL-1β, IL-4, IL-6, IL-8, IL-10, TNF-alpha, pg/mL) | Cytokine levels will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  Plasma cytokine levels at each time point, and changes from baseline
Biomarkers - Mitochondrial DNA content | mtDNA content will be compared before acupuncture and 5, 10 and 14 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 5, 10 and 14 weeks after baseline.
  Mitochondrial DNA (mtDNA) content at each time point, and changes from baseline
Biomarkers - Gray matter volume | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - White matter volume | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - Mean diffusivity | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - Fractional anisotropy | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - Radial diffusivities | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - Axial diffusivities | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Biomarkers - Resting state functional connectivities | Neuroimaging measures will be compared before acupuncture and 10 weeks after baseline for EA and sham-EA control groups. The changes will also be compared between the EA and sham-EA control groups at 10 weeks after baseline.
  Neuroimaging scans (rsfMRI, FLAIR, diffusion weighed, T1-weighted and T2-weighted sequences)
Feasibility - Recruitment (number of participants recruited) | Through study completion, approximately 2 years.
  The number of participants recruited (% of target recruitment)
Feasibility - Recruitment (rate of recruitment) | Through study completion, approximately 2 years.
  Number of patients recruited per month
Feasibility - Recruitment (reasons for declining participation) | Through study completion, approximately 2 years.
  Reasons for declining participation will be documented.
Feasibility - Recruitment (time spent on recruitment) | Through study completion, approximately 2 years.
  Time spent on recruitment, in minutes, wil be documented to assess recruitment productivity.
Feasibility - Compliance (number of acupuncture sessions successfully completed) | Through study completion, approximately 2 years.
  Number of acupuncture sessions successfully completed in total
Feasibility - Compliance (proportion of participants completing the scheduled acupuncture sessions) | Through study completion, approximately 2 years.
  Proportion of participants completing all the scheduled acupuncture sessions
Feasibility - Acceptability | Upon completion of treatment, at 10 weeks from baseline.
  Study participants will complete a questionnaire evaluating their perceptions towards the EA treatment at the end of treatment.
Feasibility - Satisfaction | Upon completion of treatment, at 10 weeks from baseline.
  Participants will be asked if they are satisfied and benefited from the treatment, and whether they would consider undergoing treatment again outside of a trial setting.
Feasibility - Blinding assessment | Upon completion of treatment, at 10 weeks from baseline.
  Participants will be asked whether they believe that they have received EA or sham-EA at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, PharmD, Principal Investigator — UCI
Locations (1):
- UCI Health Susan Samueli Integrative Health Institute, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janelsins MC, Heckler CE, Peppone LJ, Kamen C, Mustian KM, Mohile SG, Magnuson A, Kleckner IR, Guido JJ, Young KL, Conlin AK, Weiselberg LR, Mitchell JW, Ambrosone CA, Ahles TA, Morrow GR. Cognitive Complaints in Survivors of Breast Cancer After Chemotherapy Compared With Age-Matched Controls: An Analysis From a Nationwide, Multicenter, Prospective Longitudinal Study. J Clin Oncol. 2017 Feb 10;35(5):506-514. doi: 10.1200/JCO.2016.68.5826. Epub 2016 Dec 28. PMID 28029304
- [Background] Ng T, Dorajoo SR, Cheung YT, Lam YC, Yeo HL, Shwe M, Gan YX, Foo KM, Loh WK, Koo SL, Jain A, Lee GE, Dent R, Yap YS, Ng R, Chan A. Distinct and heterogeneous trajectories of self-perceived cognitive impairment among Asian breast cancer survivors. Psychooncology. 2018 Apr;27(4):1185-1192. doi: 10.1002/pon.4635. Epub 2018 Feb 1. PMID 29315963
- [Background] Cheung YT, Ng T, Shwe M, Ho HK, Foo KM, Cham MT, Lee JA, Fan G, Tan YP, Yong WS, Madhukumar P, Loo SK, Ang SF, Wong M, Chay WY, Ooi WS, Dent RA, Yap YS, Ng R, Chan A. Association of proinflammatory cytokines and chemotherapy-associated cognitive impairment in breast cancer patients: a multi-centered, prospective, cohort study. Ann Oncol. 2015 Jul;26(7):1446-51. doi: 10.1093/annonc/mdv206. Epub 2015 Apr 28. PMID 25922060
- [Background] Toh YL, Tan CJ, Yeo AHL, Shwe M, Ho HK, Gan YX, Foo KM, Chu P, Olson K, Chan A. Association of plasma leptin, pro-inflammatory adipokines and cancer-related fatigue in early-stage breast cancer patients: A prospective cohort study. J Cell Mol Med. 2019 Jun;23(6):4281-4289. doi: 10.1111/jcmm.14319. Epub 2019 Apr 23. PMID 31016867
- [Background] Cheung YT, Shwe M, Chui WK, Chay WY, Ang SF, Dent RA, Yap YS, Lo SK, Ng RC, Chan A. Effects of chemotherapy and psychosocial distress on perceived cognitive disturbances in Asian breast cancer patients. Ann Pharmacother. 2012 Dec;46(12):1645-55. doi: 10.1345/aph.1R408. Epub 2012 Dec 18. PMID 23249868
- [Background] Liou KT, Root JC, Garland SN, Green J, Li Y, Li QS, Kantoff PW, Ahles TA, Mao JJ. Effects of acupuncture versus cognitive behavioral therapy on cognitive function in cancer survivors with insomnia: A secondary analysis of a randomized clinical trial. Cancer. 2020 Jul 1;126(13):3042-3052. doi: 10.1002/cncr.32847. Epub 2020 Apr 22. PMID 32320061
- [Background] Zhang ZJ, Man SC, Yam LL, Yiu CY, Leung RC, Qin ZS, Chan KS, Lee VHF, Kwong A, Yeung WF, So WKW, Ho LM, Dong YY. Electroacupuncture trigeminal nerve stimulation plus body acupuncture for chemotherapy-induced cognitive impairment in breast cancer patients: An assessor-participant blinded, randomized controlled trial. Brain Behav Immun. 2020 Aug;88:88-96. doi: 10.1016/j.bbi.2020.04.035. Epub 2020 Apr 16. PMID 32305573
- [Background] Tong T, Pei C, Chen J, Lv Q, Zhang F, Cheng Z. Efficacy of Acupuncture Therapy for Chemotherapy-Related Cognitive Impairment in Breast Cancer Patients. Med Sci Monit. 2018 May 8;24:2919-2927. doi: 10.12659/MSM.909712. PMID 29735975
- [Background] Zeng Y, Cheng ASK, Song T, Sheng X, Wang S, Xie J, Chan CCH. Effects of Acupuncture on Cancer-Related Cognitive Impairment in Chinese Gynecological Cancer Patients: A Pilot Cohort Study. Integr Cancer Ther. 2018 Sep;17(3):737-746. doi: 10.1177/1534735418777109. Epub 2018 May 26. PMID 29806502
- [Derived] Xie L, Ng DQ, Heshmatipour M, Acharya M, Coluzzi P, Guerrero N, Lee S, Malik S, Parajuli R, Stark C, Tain R, Zabokrtsky K, Torno L, Chan A. Electroacupuncture for the management of symptom clusters in cancer patients and survivors (EAST). BMC Complement Med Ther. 2023 Mar 27;23(1):92. doi: 10.1186/s12906-023-03926-9. PMID 36973688

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT05283577/Prot_SAP_001.pdf